CLINICAL TRIAL: NCT01498198
Title: A Randomized Study of Non-Operative Management Versus Expedited Surgery Among WCB Patients With Small Rotator Cuff Tears: Affect Upon Time to Claim Closure in 2 Prairie Provinces
Brief Title: Workers Compensation Board: Rotator Cuff Tear Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Principal Investigator, Dr. Peter MacDonald, Pan Am Clinic Medical Director and University of Manitoba Faculty of Medicine Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2011:117
Record Dates: First submitted 2011-12-19; First posted 2011-12-23 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator Cuff; WCB
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expedited Surgery (Experimental): Participants will have surgery within 3 months
  Interventions: Procedure: Rotator Cuff Repair Surgery
- Non Operative Management (Experimental): Participants will undergo non operative care for as long as they are improving, and will return to the surgeon when no progression is reached.
  Interventions: Other: Non Operative Treatment

INTERVENTIONS:
Procedure: Rotator Cuff Repair Surgery — Participants will have surgery within 3 months. They will be followed up at 6 weeks, 12 weeks, 6 months and 12 months pos operatively.
  Arms: Expedited Surgery
Other: Non Operative Treatment — Participants will undergo a 6 week assessment, and if they are improving they will continue undergoing non operative care up until 12 months. If at any assessment point (6 weeks, 12 weeks, 6 months, 12 months) they are deemed to not be making any more progression, they will be referred back to the surgeon.
  Arms: Non Operative Management

SUMMARY:
The overall goal of this proposed randomized study is to determine if surgery at the time of diagnosis or rehabilitation +/- surgery (i.e. surgery only when rehabilitation fails) results in shorter times to claim closure. The study will examine how often non-operative management is successful in resolving symptoms and allowing subjects to return to work without surgery. The investigators will also examine if there are subject, tear or work-related characteristics that affect the outcome of rehabilitation or expedited surgery and predict whether patients should be referred to operative or non-operative management at time of assessment. At study completion, the investigators expect to be able to definitively state the best management for subjects with these less serious RC tears.

The specific research questions to be addressed are as follows:

1. In WCB subjects with high grade partial thickness (>50%) or small full thickness (≤ 1 cm.) rotator cuff tears, how does non-operative management (i.e. rehabilitation) or expedited surgery affect time to claim closure?
2. Are there subject, tear or work-related characteristics that affect which patient management approach will be most effective and efficient?

DETAILED DESCRIPTION:
Design/Setting The present study will be a multi-center prospective, randomized controlled trial examining WCB patients presenting to Orthopaedic specialists for RC pathology.

Selection Criteria

Adult patients with an active WCB claim, presenting with a confirmed high-grade (>50%) partial-thickness or small (≤1cm) full-thickness RC tear, will be eligible for the study. Informed consent will be attained from WCB patients attending orthopaedic clinics in the Greater Edmonton and Greater Winnipeg areas. The complete list of inclusion/exclusion criteria is as follows:

Inclusion Criteria:

1. Patient is over 18 years of age
2. Patient has an active WCB Claim
3. Patient has a high-grade (>50%) partial-thickness or small (<1cm) full-thickness tear of the supraspinatus and/or infraspinatus, as confirmed by appropriate diagnostic imaging (MRI, Arthrogram, Ultrasound)

Exclusion Criteria:

1. Patient has a full-thickness tear of the subscapularis and/or teres minor
2. Patient has a low-grade (<50%) partial-thickness tear of the supraspinatus/infraspinatus
3. Patient has a moderate to large (>1cm) full-thickness tear of the supraspinatus/infraspinatus
4. Patient has undergone previous RC surgery to the affected shoulder
5. Patient has major joint trauma, infection, or avascular necrosis
6. Patient has chronic dislocation, inflammation, or degenerative glenohumeral arthropathy
7. Patient has evidence of significant cuff arthropathy (superior glenohumeral translation and/or acromial erosion, as diagnosed by diagnostic imaging)
8. Patient has a psychiatric illness, cognitive impairment, or other health condition (i.e. visual impairment) which precludes informed consent or renders the patient unable to complete study questionnaires
9. Patient has a major medical illness where life expectancy is less than 2 years
10. Patient does not speak/read/understand English
11. Patient has no fixed address or means of contact
12. Patient unwilling to complete necessary follow-ups

Enrollment Procedures Immediately following orthopedic consultation or consultation with a screening physician, the patient will be introduced to the study. If the patient expresses interest, the Research Coordinator will discuss the study in detail (goals, requirements of patients, expected outcomes, benefits, risks) with the patient. Informed consent will be obtained from interested patients. It is expected that the patient will see the orthopaedic surgeon within three-six months of the initial presenting incident.

Baseline Evaluation Consented patients will undergo a pre-operative assessment by a study physical therapist. The assessment will consist of 1) shoulder ROM, 2) shoulder strength using a handheld myometer (microFET3, Hoggan Health Industries Inc., West Jordan, UT), 3) demographic (age, gender, height, weight, handedness, smoking status, recreational sports, date of injury, mechanism of injury) data, and 4) work-related questions (i.e. occupation, employment status, type of work performed). The subject will also complete the Western Ontario Rotator Cuff (WORC) Index.

Randomization Upon completion of the baseline assessment (to ensure blinding), patients will randomized to one of two study groups. Randomization will be stratified by type of tear (full vs. partial thickness), and by surgeon.

Patients in Group A (non-operative) will be referred to physical therapy (PT). Patients in Group B (expedited surgery) will be booked for surgery, to be completed as soon as possible (within 3 months).

Intervention Group A (non-operative) will complete a standardized PT regime. The therapy program recommended by WCB in Winnipeg will be followed and compliance with the program will be monitored. Typically, it will consist of ROM, strengthening, scapular stabilization and functional exercises, as well as pain control modalities and manual therapy techniques, as appropriate. Assessments will take place weekly by the treating therapist.

If subjects show no sign of progression, the rehabilitation regimen will stop at 6 weeks and subjects will return to the orthopaedic surgeon for a discussion of further treatment options, including surgery.

No progression will be determined by the following: the subject's total WORC score has changed less than 10% from previous assessment(baseline) and the treating PT indicates that the shoulder has not improved or worsened (using a global rating of change questionnaire - See attached document).

If subjects have made progress in PT, treatment will continue for an additional 4-6 weeks with weekly assessments of progress. PT can continue for as long as indicated, including after subject's return to work.

If at any time, the subject is determined to have stopped progressing in PT (based on comparison to previous visit) and require further evaluation, he/her will return the orthopaedic surgeon for a discussion of further options including surgery.

Group B (expedited surgery) will receive rotator cuff repair surgery. At the time of surgery, the attending surgeon will record the RC defect and repair details using a standardized form.

Follow-up Evaluations Group A1- Effective Non-operative Management: Research re-assessments will be conducted by a study physical therapist at 6 and 12 weeks, and again at 6 and 12 months after commencing PT. These re-assessments will repeat the measurements taken at the baseline evaluation and will also include a form on return to work status.

Group A2- Failed Non-operative Management: If the subjects in the non-operative group fail to progress at any point in the PT program, they will return to the orthopaedic surgeon for discussion of further treatment options, including surgery. Re-assessments will occur at the same intervals as Group A1 until such time as they receive surgery (if within the initial 12-month follow-up).

If these candidates are deemed operative and undergo surgery, they will then be followed at the same postoperative intervals as the expedited surgery group (namely 6 and 12weeks and again at 6 and 12 months postoperatively) However, the postoperative follow-up on subjects who cross over to the surgery group from the non-operative group may be less than 12 months as the study will stop when the last expedited surgery subject has reached 12 months postoperative to prevent delays in completing the study).

Group B- Expedited Surgery: Research re-assessments will be conducted by a study physical therapist at 6 and 12 weeks, and again at 6 and 12 months postoperatively. At 6 and 12 weeks, only ROM and the WORC score will be completed as well as their work status. At 6 and 12 months postoperatively, the re-assessments will repeat all measurements taken at the baseline evaluation and will also include a form on return to work status.

Outcomes The primary outcome in the present study will be time to return to final work status. The secondary outcome will be time to return to any work status (i.e. modified duties). Finally, we will also evaluate the characteristics (demographic, tear-, and work-related, ROM and strength, self-efficacy) associated with a successful outcomes among patients in both groups.

The overall goal of the study is to determine whether PT followed by surgery or expedited surgery result in a faster return to work after injury and which of these approaches are associated with the best patient outcomes within 12-months. We also hope to identify if there are sub-groups for which one approach is more effective than the other to allow optimal delivery of care.

Outcome Measures Time to Return to Work To answer our primary research question, time to return to work (in days) will be calculated. This will be defined as the interval from the date of orthopedic consultation/screening to final return to work status. We will also determine the time to any return to work status.

Demographics At each patient's pre-operative (baseline) assessment, a complete list of demographic information will be recorded. These include the patient's contact information, age, gender, height, weight, handedness, smoking status, date of injury, injury mechanism, occupation, employment status, type of work performed, and any recreational sports (type/frequency) competing in. Patients will also be asked about the particulars of any previous physical therapy regimen (where, start/stop dates, how many sessions attended), as well as any other non-operative treatments (cortisone, massage therapy, chiropractic, acupuncture).

Range of Motion Range of motion (ROM) assessments will be conducted by the study physical therapist and will performed for shoulder flexion, abduction, external rotation (neutral abduction, 90° elbow flexion), external rotation (90° abduction, 90° elbow flexion), and internal rotation (90° abduction, 90° elbow flexion). Active and passive ROM will be measured for both the operative and unaffected shoulder. ROM values will be expressed as raw values, as well as percentage of ROM compared to the unaffected shoulder.

Strength Strength assessments will also be conducted by the study physical therapist at the baseline, 6-month, and 12-month intervals. Isometric shoulder flexion, abduction, external rotation and internal rotation will be measured with the patient's arm in neutral (neutral abduction, 90° elbow flexion). Strength will be measured using a dynamometer. Peak values will be recorded during each contraction, to be held for 3 seconds each. Strength values will be expressed as raw values, as well as percentage of strength compared to the unaffected shoulder.

WORC Index The Western Ontario Rotator Cuff Index (WORC)[9] is a five-part (physical symptoms, sports/recreation, work, lifestyle, emotions), 21-item, disease-specific questionnaire which assesses quality of life among patients with RC pathology. This index has been shown to be valid, reliable and responsive in the rotator cuff patient population.

Orebro Musculoskeletal Pain Questionnaire The Orebro Musculoskeletal Pain Questionnaire (OMPQ) is a validated instrument that examines subject's ability to manage their pain during daily life. It is predictive of the subject's ability to return to work following injury and will be used at the initial assessment.

Sample Size Calculation Currently, mean WCB claim duration for Albertan RC patients is approximately 9 months (270 days) [8]. In order to have statistical power of 85% and to detect a 10% difference in this outcome (deemed clinically important to the WCB and its stakeholders) [8] between groups (s=49 days; a=0.05; b=0.15), 60 patients will be required per group. In order to allow for subject attrition, patients who may not complete all assessments due to early WCB claim closure, and to allow adequate power for subsequent multivariate regression modeling, a 20% over-sample rate will be applied. Therefore, a total of 132 patients will be recruited (66 per group) [9].

Data Analysis All study data will come from primary sources (patient assessments, surgical report forms, date of return to work at modified or full work status).

Descriptive statistics (frequency, mean, standard deviation) will be calculated for all study variables. Level of statistical significance will be set at α=0.05. All analyses will be performed using Statistical Packages for the Social Sciences (SPSS), version 16.0 (SPSS Inc.; Chicago, IL).

Three different analyses will take place. The first analysis, to address the primary research question, will count the days from screening/orthopaedic surgeon consultation to return to final work status (e.g can be either full or modified duties). In this analysis, subjects in the non-operative group will be considered as 1 group regardless of whether or not they eventually undergo surgery. If subjects have not yet returned to work when the study is deemed completed, they will be given the maximum span of days in the study (i.e. from entry to last date of study). This analysis will give the overall comparison of expedited surgery vs. initial non-operative management +/- surgical intervention, (which reflects the current standard of care).

The second analysis will look at what proportion of subjects 'fail' non-operative management. In this analysis, we will also try to identify what characteristics are associated with successful non-operative management vs. failed non-operative management.

The third analysis will examine outcomes amongst those who had successful non-operative management, those who received expedited surgery and those who underwent initial non-operative management followed by surgical intervention. This will allow us to determine the impact of delaying surgery on subjects' final outcome and if surgery results in different outcomes than non-operative management.

As the present project will assess human subjects, ethics approval will be obtained from the institutional Research Ethics Boards (REB) at the University of Manitoba and University of Alberta.

ELIGIBILITY:
Inclusion Criteria:

* Patient is over 18 years of age
* Patient has an active WCB Claim
* Patient has a high-grade (>50%) partial-thickness or small (<1cm) full-thickness tear of the supraspinatus and/or infraspinatus, as confirmed by appropriate diagnostic imaging (MRI, Arthrogram, Ultrasound)

Exclusion Criteria:

* Patient has a full-thickness tear of the subscapularis and/or teres minor
* Patient has a low-grade (<50%) partial-thickness tear of the supraspinatus/infraspinatus
* Patient has a moderate to large (>1cm) full-thickness tear of the supraspinatus/infraspinatus
* Patient has undergone previous RC surgery to the affected shoulder
* Patient has major joint trauma, infection, or avascular necrosis
* Patient has chronic dislocation, inflammation, or degenerative glenohumeral arthropathy
* Patient has evidence of significant cuff arthropathy (superior glenohumeral translation and/or acromial erosion, as diagnosed by diagnostic imaging)
* Patient has a psychiatric illness, cognitive impairment, or other health condition (i.e. visual impairment) which precludes informed consent or renders the patient unable to complete study questionnaires
* Patient has a major medical illness where life expectancy is less than 2 years
* Patient does not speak/read/understand English
* Patient has no fixed address or means of contact
* Patient unwilling to complete necessary follow-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Time to return to final work status | Participations followed for duration of the study, up to 1 year, until they fully return to work
  To answer our primary research question, time to return to work (in days) will be calculated. This will be defined as the interval from the date of orthopedic consultation/screening to final return to work status. We will also determine the time to any return to work status.

SECONDARY OUTCOMES:
Demographics | 1 year
  A complete list of demographic information will be recorded. These include the patient's contact information, age, gender, height, weight, handedness, smoking status, date of injury, injury mechanism, occupation, employment status, type of work performed, and any recreational sports (type/frequency) competing in. Patients will also be asked about the particulars of any previous physical therapy regimen (where, start/stop dates, how many sessions attended), as well as any other non-operative treatments (cortisone, massage therapy, chiropractic, acupuncture).
Range of Motion | 1 year
  Range of motion (ROM) assessments will be conducted by the study physical therapist and will performed for shoulder flexion, abduction, external rotation (neutral abduction, 90° elbow flexion), external rotation (90° abduction, 90° elbow flexion), and internal rotation (90° abduction, 90° elbow flexion). Active and passive ROM will be measured for both the operative and unaffected shoulder. ROM values will be expressed as raw values, as well as percentage of ROM compared to the unaffected shoulder.
WORC Questionnaire | 1 year
  The Western Ontario Rotator Cuff Index (WORC)[9] is a five-part (physical symptoms, sports/recreation, work, lifestyle, emotions), 21-item, disease-specific questionnaire which assesses quality of life among patients with RC pathology. This index has been shown to be valid, reliable and responsive in the rotator cuff patient population.
Orebro Questionnaire | 1 year
  The Orebro Musculoskeletal Pain Questionnaire (OMPQ) is a validated instrument that examines subject's ability to manage their pain during daily life. It is predictive of the subject's ability to return to work following injury and will be used at the initial assessment.
Strength | 1 year
  Strength assessments will also be conducted by the study physical therapist at the baseline, 6-month, and 12-month intervals. Isometric shoulder flexion, abduction, external rotation and internal rotation will be measured with the patient's arm in neutral (neutral abduction, 90° elbow flexion). Strength will be measured using a dynamometer. Peak values will be recorded during each contraction, to be held for 3 seconds each. Strength values will be expressed as raw values, as well as percentage of strength compared to the unaffected shoulder.

CONTACTS AND LOCATIONS:
Overall Officials: Peter B MacDonald, MD FRCSC, Principal Investigator — University of Manitoba Faculty of Medicine
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada